CLINICAL TRIAL: NCT07169734
Title: A Phase I/II, Open-label, Multicenter Study of ALE.P03 (Claudin-1 Targeted Antibody-drug Conjugate) as a Monotherapy in Adult Patients With Selected Advanced or Metastatic CLDN1+ Solid Tumors
Brief Title: A Study to Investigate ALE.P03 as Monotherapy in Adult Patients With Selected Advanced or Metastatic CLDN1+ Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alentis Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ALE.P03.01; 2025-521441-24-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-10; First posted 2025-09-12 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-09

CONDITIONS: Cervical Squamous Cell Carcinoma; Squamous Non-small-cell Lung Cancer; Colorectal Cancer; Intrahepatic Cholangiocarcinoma; Urothelial Carcinoma
Keywords: Claudin-1 Targeted Antibody-Drug Conjugate; Monotherapy; First-in-Human; Recommended Phase 2 dose; Recommended dose for expansion
MeSH Terms: conditions — Colorectal Neoplasms; Cholangiocarcinoma; Carcinoma, Transitional Cell

STUDY DESIGN:
Intervention Model Description: For Phase I recommended dose for expansion (RDE) part of the study, patients will be randomized in 1:1 ratio to identify the recommended Phase II dose (RP2D) for Phase II.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase I Dose Escalation- ALE.P03 (Experimental): Patients will receive ALE.P03 as monotherapy via intravenous infusion. The ALE.P03 will be given at an escalated dose until Maximum tolerated dose (MTD) and/or a safe recommended dose for expansion (RDE) is determined in Phase I dose escalation part of the study.
  Interventions: Drug: ALE.P03
- Phase I Dose Expansion- ALE.P03 (Experimental): Patients will receive ALE.P03 as monotherapy via intravenous infusion. The safe recommended doses of ALE.P03 will be given in Phase I dose expansion part of the study to identify recommended Phase II dose (RP2D) for Phase II.
  Interventions: Drug: ALE.P03
- Phase II- ALE.P03 (Experimental): Patients will receive ALE.P03 as monotherapy via intravenous infusion at the RP2D, or according to the dosing schedule after the dose expansion phase.
  Interventions: Drug: ALE.P03

INTERVENTIONS:
Drug: ALE.P03 — ALE.P03, will be administered by IV infusion according to the assigned arms.
  Arms: Phase I Dose Escalation- ALE.P03
Drug: ALE.P03 — ALE.P03, will be administered by IV infusion according to the assigned arms.
  Arms: Phase I Dose Expansion- ALE.P03
Drug: ALE.P03 — ALE.P03, will be administered by IV infusion according to the assigned arms.
  Arms: Phase II- ALE.P03

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetic, pharmacodynamic, preliminary anti-tumor activity, and to determine the recommended Phase II dose (RP2D) of the ALE.P03 monotherapy in adult patients with selected squamous solid tumors.

DETAILED DESCRIPTION:
This Study has a Phase I ALE.P03 monotherapy dose escalation and recommended dose for expansion (RDE) study and a Phase II study of ALE.P03 as monotherapy at RP2D in adult patients with selected advanced or metastatic Claudin-1 positive (CLDN1+) cancers.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically and cytologically metastatic confirmed advanced or metastatic colorectal cancer, intrahepatic cholangiocarcinoma, squamous non-small cell lung cancer, urothelial carcinoma, and cervical squamous cell carcinoma.
* Have documented radiological disease progression at study entry.
* Have provided tissue for CLDN1 (Claudin-1) analysis in a central laboratory.

Phase I Dose Escalation:

- Received and being refractory/intolerant to available systemic standard of care (SOC) regimens (based on local institutional guidelines) for advanced disease.

Phase I RDE and Phase II:

* Received 1-2 available systemic SOC regimens (based on local institutional guidelines) for advanced disease and being refractory or intolerant to treatment.
* Patients with actionable oncogenic drivers: received feasible targeted therapy.

Applicable for Phase I Dose Escalation, Phase I RDE and Phase II:

* Measurable disease per RECIST 1.1, as determined by the site.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Groups Performance Status.
* Demonstrate adequate bone marrow and organ function as per the protocol.

Exclusion Criteria:

* SqNSCLC and CSCC: diagnosed with a tumor of predominantly non-squamous histology result or adenocarcinoma.
* Has received antineoplastic therapies prior to study intervention within specified time frame.
* Has rapidly progressing disease.
* Has known active central nervous system metastases and/or carcinomatous meningitis.
* Has a history of (non-infectious) interstitial lung disease/pneumonitis that required steroids or current symptomatic or clinically significant pneumonitis requiring steroids and/or immunosuppressive therapies.
* Has clinically significant gastrointestinal bleeding.
* Has an active infection requiring systemic treatment.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2029-04-05 (Estimated); Study Completion 2029-10-04 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Dose Limiting Toxicities (DLTs) (Phase I) | Up to 28 days
  DLTs as defined in the protocol will be assessed to evaluate safety and tolerability of ALE.P03 (Phase I Dose Escalation), and to establish RP2D for ALE.P03 (Phase I RDE).
Number of Patients with Adverse Events (Phase I) | From Day 1 up to Safety follow-up (30 ± 5 days post last dose [Up to 4 years])
  Adverse events will be assessed to evaluate safety and tolerability of ALE.P03 (Phase I Dose Escalation), and to establish RP2D for ALE.P03 (Phase I RDE).
Overall Response Rate (ORR) (Phase I) | From ALE.P03 treatment initiation until at or prior to initiation of the use of new anti-cancer therapy (Up to 4 years)
  The ORR is the proportion of patients with a best overall response (BOR) of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1.) This is assessed to establish RP2D for ALE.P03 (Phase I RDE)
Duration of Response (DoR) (Phase I) | From ALE.P03 treatment initiation until disease progression or study completion (Up to 4 years)
  The DoR is defined for patients achieving a CR or PR as per Investigator review according to RECIST 1.1 to disease progression before new anti-cancer therapy or death of any cause, whichever occurs earlier. This is assessed to establish RP2D for ALE.P03 (Phase I RDE).
Overall Response Rate (ORR) (Phase II) | From ALE.P03 treatment initiation until at or prior to initiation of the use of new anti-cancer therapy (Up to 4 years)
  The ORR is assessed to assess anti-tumor activity of ALE.P03 (Phase II).
Duration of Response (DoR) (Phase II) | From ALE.P03 treatment initiation until disease progression or study completion (Up to 4 years)
  The DoR is defined for patients achieving a confirmed CR or PR as the time from the initial response of CR or PR to disease progression before new anti-cancer therapy or death of any cause, whichever occurs earlier. This is assessed to assess anti-tumor activity of ALE.P03 (Phase II).

SECONDARY OUTCOMES:
Number of Patients with Adverse Events (Phase I RDE and Phase II) | From Day 1 up to Safety follow-up (30 ± 5 days post last dose [Up to 4 years]
  Adverse events will be assessed to evaluate safety and tolerability of ALE.P03 (Phase I RDE and Phase II)
Disease control rate (DCR) (Phase I and II) | From ALE.P03 treatment initiation until at or prior to initiation of the use of new anti-cancer therapy (Up to 4 years)
  The DCR is defined as the proportion of patients with a BOR of CR or PR or stable disease (SD) per Investigator review according to RECIST 1.1 at or prior to initiation of the use of new anti-cancer therapy. This is assessed to evaluate preliminary evidence of anti-tumor activity of ALE.P03 (Phase I and II).
Median Progression-Free Survival (PFS) rate at 6 and 12 Months (Phase I and II) | At 6 and 12 months after initiation of ALE.P03 treatment
  The PFS is defined as time from first study treatment to a documented disease progression according to RECIST 1.1, as determined by the Investigator, or death due to any cause, whichever occurs earlier. This is assessed to evaluate preliminary evidence of anti-tumor activity of ALE.P03 (Phase I and II).
Median Overall Survival (OS) rate at 6, 12, and 24 Months (Phase I and II) | At 6, 12, and 24 months after initiation of ALE.P03 treatment
  The OS is defined as time from first study treatment to death due to any cause. This is assessed to evaluate preliminary evidence of anti-tumor activity of ALE.P03 (Phase I and II).
Blood Concentration of ALE.P03 Antibody-drug Conjugate (ADC) (Phase I and II) | Phase I and II: From Day 1 until at end of treatment visit (EoT) (Up to 4 years)
  Concentrations of ALE.P03 ADC in blood will be measured at each scheduled time point per arms.
Blood Concentrations of Total Antibody (Phase I and II) | Phase I and II: From Day 1 until at EoT (Up to 4 years)
  Concentrations of total antibody in blood will be measured at each scheduled time point per arms.
Blood Concentrations of Payload (Phase I and II) | Phase I and II: From Day 1 until at EoT (Up to 4 years)
  Concentrations of payload in blood will be measured at each scheduled time point per arms.
Area under the concentration-time curve over the dosing interval (AUCtau) (Phase I and II) | Phase I and II: From Day 1 until at EoT (Up to 4 years)
  The AUCtau of ALE.P03 will be measured to assess the pharmacokinetic (PK) profile of ALE.P03.
Area under the concentration-time curve from pre-dose (time 0) to the time of the last quantifiable concentration (AUClast) (Phase I and II) | Phase I and II: From Day 1 until at EoT (Up to 4 years)
  The AUClast of ALE.P03 will be measured to assess the PK profile of ALE.P03.
Area under the concentration-time curve from pre-dose (time 0) extrapolated to infinite time (AUCinf) (Phase I and II) | Phase I and II: From Day 1 until at EoT (Up to 4 years)
  The AUCinf of ALE.P03 will be measured to assess the PK profile of ALE.P03.
Maximum Concentration (Cmax) (Phase I and II) | Phase I and II: From Day 1 until at EoT (Up to 4 years)
  The Cmax of ALE.P03 will be measured to assess the PK profile of ALE.P03. It is determined directly from the concentration-time profile.
Minimum concentration (Cmin) (Phase I and II) | Phase I and II: From Day 1 until at EoT (Up to 4 years)
  The Cmin of ALE.P03 will be measured to assess the PK profile of ALE.P03. It is determined directly from the concentration-time profile.
Concentration at the end of a dosing interval (Ctrough) (Phase I and II) | Phase I and II: From Day 1 until at EoT (Up to 4 years)
  The Ctrough of ALE.P03 will be measured to assess the PK profile of ALE.P03.
The terminal elimination rate constant (KeL) (Phase I and II) | Phase I and II: From Day 1 until at EoT (Up to 4 years)
  The KeL of ALE.P03 will be measured to assess the PK profile of ALE.P03. It is determined by selection of at least three data points on the terminal phase of the concentration-time curve.
Terminal elimination half-life (t½) (Phase I and II) | Phase I and II: From Day 1 until at EoT (Up to 4 years)
  The t½ of ALE.P03 will be measured to assess the PK profile of ALE.P03.
Time of Maximum Concentration (tmax) (Phase I and II) | Phase I and II: From Day 1 until at EoT (Up to 4 years)
  The tmax of ALE.P03 will be measured to assess the PK profile of ALE.P03. It is determined directly from the concentration-time profile.
Average Concentration (Cavg) (Phase I and II) | Phase I and II: From Day 1 until at EoT (Up to 4 years)
  The Cavg of ALE.P03 will be measured to assess the PK profile of ALE.P03.
Number of Patients with Presence of anti-ALE.P03 Antibodies (Phase I and II) | Phase I and II: From Day 1 until at EoT (Up to 4 years)
  Presence of anti-ALE.P03 Antibodies will be assessed to evaluate the immunogenicity of ALE.P03.
Number of Patients with Positive anti-ALE.P03 Antibodies (Phase I and II) | Phase I and II: From Day 1 until at EoT (Up to 4 years)
  Presence of anti-ALE.P03 Antibodies (positive/negative) will be assessed to evaluate the immunogenicity of ALE.P03.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Norton Cancer Institute - Norton Healthcare Pavilion, Louisville, Kentucky
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Next Oncology-Oncology, San Antonio, Texas
  - NEXT Oncology Virginia, Fairfax, Virginia
- National Cancer Centre Singapore (NCCS), Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No